CLINICAL TRIAL: NCT06560983
Title: One Year Mortality and Morbidity Outcome With Hyperglycemia Among Acute Cerebrovascular Accident Patients in Emergency Department: A Prospective Cohort Study
Brief Title: One Year Mortality and Morbidity With Hyperglycemia Among Acute Cerebrovascular Accident Patients in Emergency Department: A Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Institute of medicine, Maharagjung medical campus (Other)
Responsible Party: Principal Investigator, Bibek Rajbhandari, Medical Doctor, Institute of medicine, Maharagjung medical campus
Other Study IDs: 6-11E2
Record Dates: First submitted 2024-08-03; First posted 2024-08-19 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Diseases
Keywords: Acute Stroke; Hyperglycemia; mortality
MeSH Terms: conditions — Cardiovascular Diseases; Stroke; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute stroke with hyperglycemia: Exposed group signifies acute stroke presenting in emergency department with hyperglycemia
  Interventions: Other: The investigators are planning to do a observational cohort study, hence won't be doing any intervention.

INTERVENTIONS:
Other: The investigators are planning to do a observational cohort study, hence won't be doing any intervention. — The investigators won't be doing any intervention since this is an observational study.

SUMMARY:
The "One Year Mortality and Morbidity Outcome with Hyperglycemia among Acute Cerebrovascular Accident Patients in Emergency Department" is an extensive prospective cohort study designed to look into how hyperglycemia affects the short- and long-term outcomes of patients who present to the emergency room with acute cerebrovascular accidents (CVAs). Worldwide, cerebrovascular accidents are a major source of both death and morbidity. Research on the long-term consequences of hyperglycemia and its association with worse outcomes during the acute period of stroke is still underway. This study aims to close this information gap by investigating the relationship between the rates of immediate short- and one-year mortality rates and morbidity and hyperglycemia at the time of CVA presentation. The research design adopts a prospective cohort approach, aligning with established guidelines to ensure methodological rigor. Systematic random sampling will be employed, with a calculated sample size of 60. Patients with acute cerebrovascular accidents who are admitted to the emergency department will be a carefully chosen group for the research. The investigators will carefully gather important data, such as baseline clinical parameters, medical history, demographics, and blood glucose levels upon admission. Throughout a year, follow-up evaluations will be carried out regularly to monitor death rates and evaluate functional and neurological results in research participants using the modified Rankin score. The study will use a structured questionnaire for data collection, involving chart review and face-to-face interviews at specified intervals. Data analysis will include bivariate analysis, logistic regression, and Kaplan-Meier analysis to identify predictors of mortality and morbidity. The ultimate goal of this research is to improve patient care, prognosis, and long-term quality of life for those impacted by this critical medical condition by illuminating the prolonged effects of hyperglycemia in acute cerebrovascular accident patients and deepening our understanding of the intricate interactions between metabolic factors and stroke outcomes.

DETAILED DESCRIPTION:
The research design and methodology of this study are meticulously crafted to explore the complex interplay between acute stroke, hyperglycemia, and their impact on mortality and morbidity. This study adopts a prospective cohort design, following a systematic approach inspired by the Critical Appraisal Skills Programme (CASP) cohort study guidelines and adhering strictly to the STROBE (Strengthening the reporting of observational studies in epidemiology), reporting standards. By implementing a quantitative research method, the study aims to provide high-quality evidence through structured and transparent methodology.

The study focuses on individuals presenting with acute stroke in the Emergency Department (ED) of Tribhuvan University Teaching Hospital (TUTH). The high patient volume and the availability of advanced diagnostic tools like CT scans make TUTH's ED an ideal setting for this research. According to internal audits, TUTH's ED receives a significant number of acute stroke patients, ensuring a robust sample for the study. The study will specifically examine acute stroke patients with concurrent hyperglycemia, utilizing a systematic random sampling technique to ensure representative and unbiased selection. The sample size was calculated using proportions from previous international studies, with adjustments for potential loss to follow-up. The final sample size is set at 60 participants, evenly divided between those with hyperglycemia and those with normal glycemic levels, allowing for meaningful comparisons.

The study's dependent variables are mortality and morbidity, assessed at short-term (1 month), mid-term (3 months), and long-term (1 year) intervals. Independent variables include demographic characteristics, clinical history, and laboratory parameters. Matching based on age, sex, stroke type, and other relevant variables is essential to minimize confounding, enhancing the validity and reliability of the study's findings. Data collection will involve chart reviews for baseline characteristics and clinical history, followed by face-to-face interviews at 1 month, 3 months, and 1 year for follow-up assessments. Laboratory analyses will be conducted for blood glucose levels, and CT scans will be utilized to confirm stroke diagnoses and assess severity. Mortality will be tracked within specified time frames, while morbidity will be assessed using the Modified Rankin Score (MRS). Clinical variables such as vital signs, GCS score, and BEFAST criteria will be recorded meticulously. Hemorrhagic and ischemic strokes will be evaluated using specific criteria, including the The intracerebral hemorrhage (ICH) score and The NIH Stroke Scale/Score (NIHSS), respectively. Participants will be recruited through a systematic process at the triage registration desk, with initial assessments based on BEFAST criteria and additional clinical signs. Blood glucose levels will be measured, followed by CT imaging to confirm stroke diagnoses. This structured flow ensures the accurate identification of eligible participants and the collection of relevant data for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals exhibiting BEFAST-positive symptoms - meeting at least one of the criteria within 24 hours of symptom onset.
* Confirmation of acute stroke through CT imaging.
* Participants aged over 40 years.

Exclusion Criteria:

* Patients presenting with hypoglycemia
* Transient Ischemic Attack (TIA).
* Subdural hematoma cases.
* Subarachnoid hemorrhage cases.
* Diabetic Ketoacidosis.
* Conditions mimicking stroke symptoms (e.g., sepsis, metabolic derangement, space-occupying lesions, hepatic encephalopathy).
* History of bedridden patients.
* Acute-on-chronic stroke cases.
* Patients requiring assistance in daily activities.
* History of trauma preceding the stroke.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * Cohort: Acute Stroke Patients
  * Sampling Frame: Individuals presenting with acute stroke in the Emergency Room
  * Sampling Unit: Acute stroke patients with concurrent hyperglycemia
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Mortality outcomes among hyperglycemic patients with acute stroke in the Emergency Department. | 1, 3, and 12 months
  Outcome Measure: Mortality rate among hyperglycemic patients with acute stroke. Unit of Measure: Percentage (%) or absolute number of deaths.
Morbidity outcomes among hyperglycemic patients with acute stroke in the Emergency Department. | 1, 3, and 12 months
  Outcome Measure: Morbidity as assessed by the Modified Rankin Scale (MRS). Unit of Measure: MRS score (scale of 1 to 5).
  Morbidity Assessment: The Modified Rankin Scale (MRS) will be used to quantify the degree of functional impairment or disability resulting from the acute stroke. The MRS score ranges from 1 to 5, with 1 indicating minimal symptoms and 5 representing severe disability or bedridden status.

SECONDARY OUTCOMES:
Demographic Characteristics and Mortality Outcomes | 1, 3, and 12 months
  Outcome Measure: Mortality rate stratified by demographic characteristics (age, sex, ethnicity, socioeconomic status).
  Unit of Measure: Percentage (%) or number of deaths per group.
Type of Stroke and Mortality Outcomes | 1, 3, and 12 months
  Outcome Measure: Mortality rate stratified by type of stroke (ischemic, hemorrhagic, other). Unit of Measure: Percentage (%) or number of deaths per stroke type.
Clinical History and Mortality Outcomes | 1, 3, and 12 months
  Outcome Measure:Mortality rate stratified by clinical history (presence of comorbid conditions, previous strokes, BMI, smoking habits, alcohol consumption). Unit of Measure: Percentage (%) or number of deaths per clinical history category
Laboratory Parameters and Mortality Outcomes | 1, 3, and 12 months
  Outcome Measure: Mortality rate stratified by laboratory parameters (e.g., blood glucose levels, cholesterol levels). Unit of Measure: Percentage (%) or number of deaths per laboratory parameter range.
Treatment and Mortality Outcomes | 1, 3, and 12 months
  Outcome Measure: Mortality rate stratified by type of treatment (e.g., medications, surgical interventions). Unit of Measure: Percentage (%) or number of deaths per treatment type.

CONTACTS AND LOCATIONS:
Locations (1):
- Bibek Rajbhandari, Kathmandu, Bagmati, Nepal

REFERENCES:
- [Background] GBD 2016 Stroke Collaborators. Global, regional, and national burden of stroke, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. Lancet Neurol. 2019 May;18(5):439-458. doi: 10.1016/S1474-4422(19)30034-1. Epub 2019 Mar 11. PMID 30871944
- [Background] Bender M, Jusufovic E, Railic V, Kelava S, Tinjak S, Dzevdetbegovic D, Mot D, Tresnjo M, Lakicevic S, Pejanovic-Skobic N, Sinanovic O. High Burden of Stroke Risk Factors in Developing Country: the Case Study of Bosnia-Herzegovina. Mater Sociomed. 2017 Dec;29(4):277-279. doi: 10.5455/msm.2017.29.277-279. PMID 29284999
- [Background] Lindsay MP, Norrving B, Sacco RL, Brainin M, Hacke W, Martins S, Pandian J, Feigin V. World Stroke Organization (WSO): Global Stroke Fact Sheet 2019. Int J Stroke. 2019 Oct;14(8):806-817. doi: 10.1177/1747493019881353. No abstract available. PMID 31658892
- [Background] Pandian JD, Sudhan P. Stroke epidemiology and stroke care services in India. J Stroke. 2013 Sep;15(3):128-34. doi: 10.5853/jos.2013.15.3.128. Epub 2013 Sep 27. PMID 24396806
- [Background] Feigin VL, Lawes CM, Bennett DA, Barker-Collo SL, Parag V. Worldwide stroke incidence and early case fatality reported in 56 population-based studies: a systematic review. Lancet Neurol. 2009 Apr;8(4):355-69. doi: 10.1016/S1474-4422(09)70025-0. Epub 2009 Feb 21. PMID 19233729
- [Background] Donkor ES. Stroke in the 21st Century: A Snapshot of the Burden, Epidemiology, and Quality of Life. Stroke Res Treat. 2018 Nov 27;2018:3238165. doi: 10.1155/2018/3238165. eCollection 2018. PMID 30598741
- [Background] Bates BE, Xie D, Kwong PL, Kurichi JE, Ripley DC, Stineman MG. One-year all-cause mortality after stroke: a prediction model. PM R. 2014 Jun;6(6):473-83. doi: 10.1016/j.pmrj.2013.11.006. Epub 2013 Nov 7. PMID 24211696
- [Background] Mar J, Masjuan J, Oliva-Moreno J, Gonzalez-Rojas N, Becerra V, Casado MA, Torres C, Yebenes M, Quintana M, Alvarez-Sabin J; CONOCES Investigators Group. Outcomes measured by mortality rates, quality of life and degree of autonomy in the first year in stroke units in Spain. Health Qual Life Outcomes. 2015 Mar 17;13:36. doi: 10.1186/s12955-015-0230-8. PMID 25889480
- [Background] Liljehult J, Christensen T, Christensen KB. Early Prediction of One-Year Mortality in Ischemic and Haemorrhagic Stroke. J Stroke Cerebrovasc Dis. 2020 Apr;29(4):104667. doi: 10.1016/j.jstrokecerebrovasdis.2020.104667. Epub 2020 Feb 8. PMID 32044222
- [Background] Goulart AC, Bensenor IM, Fernandes TG, Alencar AP, Fedeli LM, Lotufo PA. Early and one-year stroke case fatality in Sao Paulo, Brazil: applying the World Health Organization's stroke STEPS. J Stroke Cerebrovasc Dis. 2012 Nov;21(8):832-8. doi: 10.1016/j.jstrokecerebrovasdis.2011.04.017. Epub 2011 Jun 25. PMID 21705233